CLINICAL TRIAL: NCT05038917
Title: Sedation for Endoscopic Procedures - a Follow-up Study of Efficiency and Safety
Brief Title: Sedation for Endoscopic Procedures
Acronym: SEEUPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Andreas Nilsson, Senior nurse anesthetist, Researcher, Principal Investigator, Ostergotland County Council, Sweden
Other Study IDs: SEEUPP 04545/02915
Record Dates: First submitted 2021-05-26; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Endoscopic Surgical Procedure
Keywords: Quality of recovery; Health Literacy; Moderate sedation; Deep sedation; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Endoscopic procedures for biliary strictures, stenting or drainage (ERCP) and ultrasonic imaging or biopsies (EUS) are performed under sedation or anesthesia. The main purpose of the study is to evaluate aspects of procedure treatability and patients´ quality of recovery.

DETAILED DESCRIPTION:
The main aim of this study is to evaluate the effects on treatability and procedure failur; also aspects of post-procedure quality of recovery from patients cognitive function and from the choice of sedation/anesthesia for ERCP and EUS-procedures.

Before endoscopic procedures, patients do not always read the written information sent to them. That´s a problem since patients tend to be insufficient prepared for the procedures. Therefore, evaluation of patients' health literacy was performed.

Patients are sedated (patient-controlled sedation or by nurse anesthetists) or in general anesthesia. No randomisation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years)
* Patients cheduled for ERCP or/and EUS
* Patients who have given their informed and written concent to participate

Exclusion Criteria:

Patients with

* confusion
* dementia
* communication problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) scheduled for ERCP or/and EUS
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Dimensions of recovery recorded by Quality of Recovery 15 swedish version | Baseline (Day 0)
  Quality of recovery (QoR15 swedish version) Max 150 points Min 0, higher scores are better
Dimensions of recovery recorded by Quality of Recovery 15 swedish version | Day 1
  Quality of recovery (QoR15 swedish version) Max 150 points Min 0, higher scores are better
Dimensions of recovery recorded by Quality of Recovery 15 swedish version | Day 5
  Quality of recovery (QoR15 swedish version) Max 150 points Min 0, higher scores are better

SECONDARY OUTCOMES:
Health literacy measured by the use of FHL (swedish version) | Before procedure (Day 0)
  Health literacy (FHL swedish version), Max 0 Min 5, 0 is good, 5 is bad
Aborted or increased difficulty to performed the planned procedure | From start of procedure to the end of it (Day 0)
  Procedure failure, numbers of aborted procedures and numbers of difficult performance

CONTACTS AND LOCATIONS:
Overall Officials: Andreas o Nilsson, PhD, Study Chair — Ljungsborg Haga 1
Locations (1):
- University hospital of Linköping, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
No sharing plans